CLINICAL TRIAL: NCT03920358
Title: FRED/ FRED Jr/ FRED X Intracranial Aneurysm Treatment Study
Acronym: FRITS
Status: Active, not recruiting | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP EMEA 18-01
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FRED, FRED Jr and FRED X — Subjects aged ≥ 18 requiring treatment for an unruptured or recanalized intracranial aneurysm
  Other Names: Flow Re-Direction Endoluminal Device

SUMMARY:
A prospective, multicenter, observational evaluation of the safety and efficacy of the FRED® device in the treatment of intracranial aneurysms

DETAILED DESCRIPTION:
This is a multi-center observational study. Treatment and follow-up visits will be performed as per standard of care. The purpose of this study is to demonstrate that use of the FRED/ FRED Jr/ FRED X Embolic device in intracranial aneurysm treatment is safe and effective when assessed at 6, 12 months and yearly up to 5 years post procedure.

150 patients will be enrolled over an 15-month recruitment period. All patients will be followed for 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years old
2. Patient harboring a non-acutely ruptured intracranial aneurysm within the last 30 days of presentation:

   * for which use of FRED, FRED Jr or FRED X has been deemed appropriate
   * being the only aneurysm to require treatment within the next 12 months
   * and optionally previously treated by surgery (clipping) or with an intrasaccular device: aneurysm recanalized
3. Patient with a modified Rankin Scale (mRS) ≤ 2
4. Patient has received information about data collection and has signed and dated an Informed Consent Form

Exclusion Criteria:

1. Patient has suffered from an ICH within the 30 days prior to the procedure.
2. The aneurysm to be treated is associated with a cAVM
3. The aneurysm to be treated is in the posterior circulation
4. The aneurysm to be treated has a stenosis of its parent artery >50%
5. Patient has another aneurysm previously treated with a stent or a flow diverter

   * on the same parent vessel at any time
   * on a different parent vessel, less than 3 months prior to the procedure (previously-implanted stents in the non-index proximal carotid are acceptable)
6. Patient with whom anticoagulant, antiplatelet or thrombolytic drugs are contra-indicated or test performed regarding AP medication administered is not efficient for the patient
7. Patient with known hypersensitivity to contrast products or nickel titanium, not treatable
8. Pregnancy or child breastfeeding
9. Patient unable or unlikely to complete required follow up
10. Patient has severe or fatal comorbidity or a life expectancy of less than 1 year
11. Treatment with a flow diverter other than FRED/ FRED Jr/ FRED X or in addition to FRED/ FRED Jr/ FRED X is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 18 years of age presenting with an unruptured or recanalized intracranial aneurysm requiring endovascular treatment. Those eligible to be treated with FRED/ FRED Jr/ FRED X will be enrolled after having signed an informed consent form.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete aneurysm occlusion without associated stenosis of the parent artery (> 50%) | 12 months
  Complete occlusion (Raymond Scale grade I) without stenosis of the parent artery.
  Raymond scale definition: Grade I= complete occlusion of aneurysm, Grade II= Residual neck, Grade III= Residual aneurysm
Morbidity Rate | 6 months
  Patients with mRS>2
Mortality Rate | 6 months
  Deaths within 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Dörfler, Prof. Dr. med., Principal Investigator — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No